CLINICAL TRIAL: NCT05566626
Title: A Single Centre, Controlled, Investigation to Evaluate the Performance of the Hyperspectral Camera for Retinal Non-invasive Examination Through the Observation of Retinal Oxygenation
Brief Title: Retinal Oxygenation Estimation Trial With Mantis Photonics Hyperspectral Camera
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Mantis Photonics AB (Industry)
Collaborators: Sundets Ögonläkare (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MANTIS_2022_08_Oxygenation_S
Record Dates: First submitted 2022-09-22; First posted 2022-10-04 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Glaucoma Eye; Macular Degeneration; Macula Abnormality; Retinal Detachment
Keywords: hyperspectral; retinoscopy; oxygenation; non-invasive
MeSH Terms: conditions — Macular Degeneration; Retinal Detachment

STUDY DESIGN:
Intervention Model Description: Alle participants, both healthy subjects and patients, receive the same intervention: hyperspectral image with Mantis Photonics camera
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camera test group (Experimental): The Principal Investigator will take a hyperspectral image of all subjects, both healthy volunteers and patients.
  Interventions: Device: Hyperspectral retinal image; Drug: Mydriacyl Ophthalmic Product

INTERVENTIONS:
Device: Hyperspectral retinal image — Hyperspectral image of both eyes
  Other Names: hyperspectral retinoscopy
Drug: Mydriacyl Ophthalmic Product — Mydriatic drops before retinoscopy

SUMMARY:
An explorative study of the Mantis Photonics hyperspectral camera for retinal imaging and estimation of retinal oxygenation.

Primary objective: To evaluate the performance of the hyperspectral camera for non-invasive retinal examination in order to improve the diagnosis of diseases affecting the retina or central nervous system. Secondary objective: To investigate the possibilities of the use of a hyperspectral camera for non-invasive retinal examination.

DETAILED DESCRIPTION:
In the retina, light is captured and then transported via the optic nerve to the brain. Common diseases in the retina are glaucoma, diabetes and age-related changes in the macular area. Diagnosing these diseases is important to be able to treat them in time. Currently, it is possible to image the retina with, for example, a regular camera or with ultrasound. Similarly, with Optical Coherence Tomography (OCT) one can get a deep view of the layers of the retina. It is currently difficult to investigate the oxygenation level of the retina. With intravenous injection followed by photography, images can be collected of the retina that shows areas of non-perfusion. However, injecting a drug is not always possible and is also associated with risk.

Mantis Photonics AB has developed a new diagnostic camera that uses an ordinary camera's light flash but analyses the reflected light with a novel patented technology into different wavelengths allowing hyperspectral imaging (HI). With HI it is possible to capture and see changes that are not visible with a regular camera. Interpretation of the reflected spectrum allows assessment of retinal oxygenation. The oxygenation level is affected in several retinal diseases, such as diabetes and glaucoma. Initial reports have shown that the technology could be valuable for early detection of, for example, diabetic retinopathy. Furthermore, hyperspectral imaging can be used to detect molecular changes seen in age-related macular degeneration.

It is believed that hyperspectral technology can provide detailed information about various disease states in the retina, such as haemorrhages, ischemia, diabetes, and glaucoma. With improved examination technology, it is possible to sharpen treatment and perhaps advance adequate treatment. This project aims to investigate, explore and refine hyperspectral camera technology by photographing healthy retinas. Furthermore, the project intends to examine people with retinal diseases such as glaucoma and age-related macular changes, diabetes, retinal detachment and compare diagnostic accuracy with other available techniques.

ELIGIBILITY:
For inclusion in the investigation, the patient-subjects must fulfill all of the below criteria prior to enrollment: 1. Age > 18 years. 2. Ophthalmological disease, disorder, illness or problem involving the retina 3. Provision of informed consent i.e., subject must be able to understand and sign the patient information and consent form. For inclusion in the investigation, the healthy subjects must fulfill all of the below criteria prior to enrollment:

1. Age >18 years.
2. Without known eye disease.
3. Provision of informed consent i.e., subject must be able to understand and sign the patient information and consent form.

Patients-subjects who meet any of the below criteria will be excluded from the investigation:

1. Patients with narrow angle glaucoma
2. Inclusion in other ongoing investigations at present that would preclude the subject from participating in this investigation as judged by the Principal Investigator. Healthy subjects who meet any of the below criteria will be excluded from the investigation:

1. Presence of eye disease, eye trauma, diabetes or pregnancy. 3. Inclusion in other ongoing investigations at present that would preclude the subject from participating in this investigation as judged by the Principal Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Performance evaluation - Retinal Oxygenation | During the procedure (retinoscopy with hyperspectral camera).
  Measurement of retinal oxygenation for each patient:
  hemoglobin oxygenation of retinal artery [in percent] hemoglobin oxygenation of retinal vein [in percent]
  Measurement: calculated result based on the hyperspectral reflectance profile of vein and artery regions of the retina.

SECONDARY OUTCOMES:
Retinal examination exploration - detection of macular degeneration | After the procedure (retinoscopy with hyperspectral camera). Manual evaluation in the week after the procedure.
  Measurement:
  Evaluation of spatial uniformity of spectral images. Observation of 'spots' and features apart from vascular features and optical nerve in single-frequency slices of the hyperspectral cube (notably between 550 and 600 nm) can indicate retinal and macular degeneration before this is observable with other means.
  Measurement is the expert evaluation of the single frequency slices for abnormalities.

OTHER OUTCOMES:
Adverse effect | Immediately after the retinoscopy procedure.
  Measurement:
  Percentage of patients who report adverse effects such as transient 'imprint' of the flash or other adverse effects.
Serious adverse effect | Immediately after the retinoscopy procedure.
  Occurrence of serious adverse effects due to procedure
  Any patient who suffers serious harm due to procedure is a study outcome and a study endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Madeleine Selvander, MD, Principal Investigator — Sundets Ögonläkare
Locations (1):
- Sundets Ögonläkare, Helsingborg, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No
No Individual Participant Data (IPD) sharing to third parties. Data of individual participants will be used for this study only.

REFERENCES:
- [Background] Bernardes R, Serranho P, Lobo C. Digital ocular fundus imaging: a review. Ophthalmologica. 2011;226(4):161-81. doi: 10.1159/000329597. Epub 2011 Sep 22. PMID 21952522
- [Background] Hardarson SH, Stefansson E, Bek T. Retinal oxygen saturation changes progressively over time in diabetic retinopathy. PLoS One. 2021 May 12;16(5):e0251607. doi: 10.1371/journal.pone.0251607. eCollection 2021. PMID 33979414
- [Background] Johnson WR, Wilson DW, Fink W, Humayun M, Bearman G. Snapshot hyperspectral imaging in ophthalmology. J Biomed Opt. 2007 Jan-Feb;12(1):014036. doi: 10.1117/1.2434950. PMID 17343511
- [Background] Lee EJ, Kee HJ, Han JC, Kee C. Evidence-based understanding of disc hemorrhage in glaucoma. Surv Ophthalmol. 2021 May-Jun;66(3):412-422. doi: 10.1016/j.survophthal.2020.09.001. Epub 2020 Sep 17. PMID 32949554
- [Background] Lu G, Fei B. Medical hyperspectral imaging: a review. J Biomed Opt. 2014 Jan;19(1):10901. doi: 10.1117/1.JBO.19.1.010901. PMID 24441941
- [Background] Meinke M, Muller G, Helfmann J, Friebel M. Empirical model functions to calculate hematocrit-dependent optical properties of human blood. Appl Opt. 2007 Apr 1;46(10):1742-53. doi: 10.1364/ao.46.001742. PMID 17356617
- [Background] Ohno-Matsui K. Parallel findings in age-related macular degeneration and Alzheimer's disease. Prog Retin Eye Res. 2011 Jul;30(4):217-38. doi: 10.1016/j.preteyeres.2011.02.004. Epub 2011 Mar 25. PMID 21440663
- [Background] Safi H, Safi S, Hafezi-Moghadam A, Ahmadieh H. Early detection of diabetic retinopathy. Surv Ophthalmol. 2018 Sep-Oct;63(5):601-608. doi: 10.1016/j.survophthal.2018.04.003. Epub 2018 Apr 19. PMID 29679616

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-10): https://cdn.clinicaltrials.gov/large-docs/26/NCT05566626/Prot_SAP_000.pdf